CLINICAL TRIAL: NCT03280043
Title: Does Ketorolac Increase the Risk of Hematoma After Reduction Mammoplasty? A Case-control Study.
Brief Title: Risk of Hematoma After Ketorolac Use in Reduction Mammoplasty.
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 1094-C
Record Dates: First submitted 2017-05-24; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Reduction; Reduction Mammoplasty; Hematoma; Hemorrhage
Keywords: Breast reduction; Reduction mammoplasty; Hematoma; Hemorrhage; Ketorolac; Toradol
MeSH Terms: conditions — Hematoma; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Women who underwent reduction mammoplasty and then developed a hematoma which required return to the operating room for evacuation.
  Interventions: Procedure: Hematoma
- Controls: Women who had uncomplicated reduction mammoplasty.

INTERVENTIONS:
Procedure: Hematoma — Hematoma requiring return to operating room.
  Groups: Cases

SUMMARY:
The investigators hope to answer the question, "does ketorolac increase the risk of hematoma after reduction mammoplasty?" using a case-control study. All patients who developed a hematoma post reduction mammoplasty (cases) at our institution, and match these with women who had an uncomplicated reduction mammoplasty (controls), and then compare frequency of ketorolac exposure between these two groups as the primary outcome. If ketorolac increases the risk of hematoma, one should expect cases to have been exposed to ketorolac more frequently than controls. Based on previously existing literature, the investigators hypothesize that cases and controls will not differ in their ketorolac exposure, that is, ketorolac does not increase the risk of hematoma.

DETAILED DESCRIPTION:
The electronic health record databases of St. Joseph's Healthcare Hamilton and Hamilton Health Sciences will be searched, using the coding system, for all cases of reduction mammoplasty with post--operative hematoma as a complication. Only hematomas which required return to the operating room for evacuation will be included (i.e. those treated with observation or needle aspiration will be excluded).

Cases are defined as patients suffering a hematoma post reduction mammoplasty will be identified through hospital coding, and matched with controls based on the following criteria: age, body mass index (BMI), pre-existing hypertension, and institution. Controls are defined as patients who had uncomplicated reduction mammoplasty, and will be randomly pulled through retrospective chart review within the same databases, in the same time period (±5 years).

All patient data will be de--identified, and all devices containing patient information will remain on hospital grounds, and be encrypted according to our hospital protocols. The following data will be extracted from patient charts: age, date of surgery, body mass index, surgeon, anesthetist, volume of breast tissue removed per breast, comorbidities, platelet count, coagulation profile, ketorolac and opioid use including dose, timing, frequency, duration, and route of administration of both, time to discharge including length of stay if overnight, comorbidities (including smoking status), American Society of Anesthesiology score, and post--operative usage of drains.

Matching of cases and controls will be performed by the primary investigator (JB), and at the time of matching, the only visible patient information will be the de-identified patient identification (ID) and the four matching variables (ketorolac exposure was not visible).

The frequency of ketorolac exposure between cases and controls will then be reviewed, and the odds ratio (OR) of exposure to ketorolac, with 95% confidence intervals will be calculated. A two by two table will be generated from our data. Since the incidence of hematoma formation after reduction mammoplasty is very low, the odds ratio will closely approximate the relative risk. To evaluate the statistical significance of the ORs, a level of significance of 0.05 will be used. Independent samples t-test will be used to compare continuous demographic data, and Chi-square analysis will be used for ordinal or categorical data between cases and controls.

Sample size was calculated using the POWER program, described by Dupont and Plummer in 1990. A sample size of 25 cases matched with 25 controls (total n = 50) was required from the following data:

* p0 = 0.32 (approximate rate of ketorolac exposure amongst breast reduction patients from previous literature from Cawthorn et al.)
* α = 0.05 (chance of type I error)
* P = 0.8 (power)
* m = 1 (matching ratio1:1)
* Ψ = 3.6 (estimated risk ratio of developing hematoma post breast reduction if exposed to ketorolac, Cawthorn et al.)
* Φ = 0.2 (measurable difference)

ELIGIBILITY:
Inclusion Criteria:

Cases:

- Patients who developed hematoma post-reduction mammoplasty requiring repeat surgery

Controls:

- Uncomplicated bilateral reduction mammoplasty

Exclusion Criteria:

* Hematoma patients treated with observation or needle aspiration
* Concomitant surgeries in addition to the reduction mammoplasty
* Allergy/sensitivity to non-steroidal anti-inflammatory drugs
* Unilateral reduction mammoplasty
* Male reduction mammoplasty
* Documented bleeding disorders

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical coders will identify all possible cases of hematoma by searching the key words "hemorrhage," "hematoma," and "plastic surgery". Hematomas post reduction mammoplasty will be manually retrieved and reviewed. Control patients will be randomly pulled from the database of uncomplicated reduction mammoplasties.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Ketorolac exposure. | Sept 2015 - Aug 2017.
  Whether or not cases and controls were exposed to ketorolac on the day of surgery will be determined and compiled as a categorical variable (yes/no).

SECONDARY OUTCOMES:
Year of reduction mammoplasty. | Sept 2015 - Aug 2017.
  The year of which the reduction mammoplasty occurred will be recorded for cases and controls. The investigators will then calculate the mean year which the reduction mammoplasty surgery occurred for the case and control groups, to ensure that on average, each group is similar in terms of the year the surgeries occurred.
Age of patients in each group will be calculated. | Sept 2015 - Aug 2017.
  Age, extracted from the medical chart, will be aggregated and mean age for cases and controls will be calculated.
Body mass index compared between cases and controls. | Sept 2015 - Aug 2017.
  BMI will be calculated for each patient from height and weight available in the medical chart, and mean BMI between case and control groups will be compared.
Volume of breast tissue resected during surgery (in grams) for each patient. | Sept 2015 - Aug 2017.
  Mean volume of breast tissue resected from each breast, which is a routinely recorded number during reduction mammoplasty, will be extracted for each patient, and mean volumes resected will be compared between cases and controls.
Pre-operative platelet count. | Sept 2015 - Aug 2017.
  Platelet counts, if available, will be extracted for each patient and means for cases and controls will be compared.
Smoking status. | Sept 2015 - Aug 2017.
  Active smokers (yes/no) will be determined by reviewing the pre-operative anesthesia records which routinely contain this information.
American society of anesthesiologist (ASA) score. | Sept 2015 - Aug 2017.
  This is an ordinal score (ASA 1 through 4) given to all patients pre-operatively, as a general indicator of risk of morbidity and mortality with a general anesthetic. This will be extracted for each patient from the pre-operative anesthesia records and frequencies of patients who are ASA 1, ASA 2, ASA 3, or ASA 4 will be aggregated and compared between cases and controls.
Specific breast side of hematoma occurrence (left versus right). | Sept 2015 - Aug 2017.
  In patients who developed a hematoma (cases), the investigators will record whether this occurred on the left, right, or both breasts.
Post-operative opioid consumption. | Sept 2015 - Aug 2017.
  The investigators will calculate post-operative opioid consumption for each patient in the study. Values will be converted to equivalence of oral morphine, in milligrams, using standard conversion charts. Mean opioid consumption will be compared between patients who received ketorolac and those who did not.
Surgeon's description of bleeding encountered during hematoma take-back. | Sept 2015 - Aug 2017.
  The investigators will review transcribed dictations of the surgeon for hematoma cases in order to determine what type of bleeding was encountered during take-back surgery. The categorical descriptors will be: pulsatile bleeding, general ooze, or both. The investigators will compare descriptors between patients who received ketorolac and those who did not.
Ketorolac dose. | Sept 2015 - Aug 2017.
  Amongst cases and controls who received ketorolac, the specific dose of ketorolac given will be recorded in milligrams.
Ketorolac route given. | Sept 2015 - Aug 2017.
  Amongst cases and controls who received ketorolac, the route which ketorolac was given will be recorded as a categorical variable (intra-venous, intra-muscular, or oral).
Timing of ketorolac dose. | Sept 2015 - Aug 2017.
  Amongst cases and controls who received ketorolac, the timing of the dose given will be recorded (i.e. pre-operative, intra-operative, or post-operative).

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD, MSc, BSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cawthorn TR, Phelan R, Davidson JS, Turner KE. Retrospective analysis of perioperative ketorolac and postoperative bleeding in reduction mammoplasty. Can J Anaesth. 2012 May;59(5):466-72. doi: 10.1007/s12630-012-9682-z. Epub 2012 Mar 21. PMID 22434401